CLINICAL TRIAL: NCT06013865
Title: An Exploratory Investigation of the Safety of Empagliflozin in Kidney Transplant Recipients (SEKTR)
Brief Title: Empagliflozin Treatment in Kidney Transplant Recipients
Acronym: SEKTR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Iowa City VA Health Care System (U.S. Federal Agency); VA Pittsburgh Healthcare System (U.S. Federal Agency); VA Tennessee Valley Health Care System (U.S. Federal Agency); VA Hines Health Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPH-008-22F; CSR&D (Other Grant/Funding Number: VHA 1 IO1 CX002666-01)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Chronic Kidney Disease
Keywords: Transplant; Diabetes; Kidney Failure; Rejection; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Renal Insufficiency; Rejection, Psychology; Proteinuria | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective Observational Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Other): Open Label, Empagliflozin 12.5 mg QD
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — SGLT2 Inhibitor
  Other Names: jardiance

SUMMARY:
Kidney transplantation improves the health and quality of life for those Veterans with end stage kidney disease (ESKD). While early patient and graft survival are excellent, long-term outcomes continue to be challenging. Patient death with existing kidney graft function occurs in about half of all recipients over time. This is primarily due to the development of cardiovascular disease in a patient population with multiple preexisting cardiac disease risk factors. There has been little progress in improving outcomes in this area for over two decades. Recent studies in chronic kidney disease (CKD) patients using SGLT2 inhibitors (SGLT2i), regardless of the presence of type 2 diabetes mellitus (T2DM), results in both kidney protective and cardiac protective impacts and improved patient outcomes. However, kidney transplant recipients (KTRs) were excluded from these clinical trials due to concerns that these agents promote infection, diminish graft function, and may alter immunosuppressive drug levels that are the mainstay of patient's transplant therapy. There are limited published data of SGLT2i treatment of selected KTRs.

DETAILED DESCRIPTION:
Background: Kidney transplantation improves the health and quality of life for those veterans with end stage kidney disease (ESKD). While early patient and graft survival are excellent, long-term outcomes continue to be challenging. Patient death with existing kidney graft function occurs in about half of all recipients over time. This is primarily due to the development of cardiovascular disease in a patient population with multiple preexisting cardiac disease risk factors. There has been little progress in improving outcomes in this area for over two decades. Recent studies in chronic kidney disease (CKD) patients using SGLT2 inhibitors (SGLT2i), regardless of the presence of type 2 diabetes mellitus (T2DM), results in both kidney protective and cardiac protective impacts and improved patient outcomes. However, kidney transplant recipients (KTRs) were excluded from these clinical trials due to concerns that these agents promote infection, diminish graft function, and may alter immunosuppressive drug levels that are the mainstay of patient's transplant therapy. There are limited published data of SGLT2i treatment of selected KTRs.

Objective: The goal of this submission is to examine the safety and efficacy of SGLT2i therapy in Veterans with KTRs with and without T2DM. The hypothesis is treatment with SGLT2i will lead to improvements in graft and cardiovascular outcomes in patients with chronic kidney disease, with acceptable side effect profile.

Methods: To test this hypothesis, the investigators will execute a multicenter clinical trial at 5 VA medical centers, including 4 that serve as primary kidney transplant programs. The multidisciplinary research team includes transplant medical and surgical expertise, diabetology, and informatics and statistical support familiar with VA data systems. In open label fashion, the investigators will treat eligible KTRs and comprehensively assess adverse and serious adverse event data, as well as assess any untoward impacts on graft function and diabetes management. Secondly, the investigators will utilize VA data from the VINCI corporate data warehouse to develop a control cohort of Veterans with KTRs with and without T2DM, not treated with SGLT2i. The investigators will utilize propensity score matching to reduce bias that may occur in observational studies. With this strategy, the investigators will further address the potential beneficial impact of SGLT2i treatment on cardiovascular outcomes, as well as kidney disease progression in the transplanted kidney. The investigators will also analyze the cost impact of using this agent in this patient population, in terms of hospitalizations, unanticipated procedures, and CKD management.

Findings: These studies will provide new information to the transplant community for both Veteran and non-Veteran alike, with a detailed assessment of safety and feasibility of this agent class using a pragmatic approach to transplant care. These results will translate into an opportunity to mitigate late graft loss in this patient population, and a potential breakthrough in clinical care that to date has been unrecognized.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years of age) male and female recipients (all races and ethnicities)
2. Subject must be able to understand and provide consent
3. Recipient of a primary or secondary kidney transplant at least 3 months or longer since transplant
4. For subjects with T2DM or post-transplant diabetes (PTDM), measured kidney function by CKD epi eGFR must be 30mL/min/1.73m2 to < 45ml/min/1.73m2 or CKD epi eGFR 45 mL/min/1.73m2 to 90ml/min/1.73m2 with urinary albumin:creatinine ratio 200 mg/g (or protein:creatinine 300 mg/g).
5. For subjects without T2DM or PTDM: measured kidney function by CKD epi eGFR must be 20mL/min/1.73m2 to < 45ml/min/1.73m2 or CKD epi eGFR 45 mL/min/1.73m2 to 90ml/min/1.73m2 with urinary albumin:creatinine ratio 200 mg/g (or protein:creatinine 300 mg/g).

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. History of prior pancreas transplant
3. CKD epi eGFR < 30 mL/min/1.73m2 for those with T2DM or < 20 mL/min/1.73m2 for those without T2DM or anyone with 5mL/min/1.73m2 fall in eGFR per year
4. Uncontrolled type 2 diabetes mellitus with most recent A1C>12%
5. History of >2 urinary tract infections per year or UTIs requiring admission in the last year, or urosepsis in the last year.
6. Use of SGLT2i within 90 days
7. Documented allergy to SGLT2i
8. History of Type I diabetes mellitus
9. History of diabetic ketoacidosis
10. Indwelling foley catheter or urinary diversion
11. Acute rejection in the prior 3 months
12. Acute MACE event within 3 months of the study
13. Severe congestive heart failure (NYHA functional class III or higher)
14. Active mucocutaneous mycotic infection of the groin or external genitalia.
15. History of amputation due to peripheral vascular disease and/or diabetic foot ulcers within prior year
16. History of malignancy except non-melanoma skin cancer within 2 years of screening
17. Known of active current viral, fungal, mycobacterial, or other infections (including, but not limited to tuberculosis and atypical mycobacterial disease)
18. HIV infected subjects, including those who are well controlled on anti-retrovirals
19. Recent (within 6 months) Positive Hep B PCR or active disease
20. Hepatitis C virus antibody positive (HCVAb+) subjects who have failed to demonstrate sustained viral remission for more than 12 weeks (after anti-viral treatment)
21. Active pregnancy in a female transplant recipient
22. A condition, in the eyes of the investigator, that precludes inclusion into the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Discontinuation of Empagliflozin | about 2 years
  The incidence of therapeutic discontinuation of empagliflozin in the kidney transplant recipient from time of initiation.

SECONDARY OUTCOMES:
Infection | about 2 years
  Defined as the cumulative incidence of study defined Grade 3 or higher infection of the urinary tract or perineum after initiation of treatment.
Hypoglycemia | about 2 years
  The cumulative incidence of grade 3 hypoglycemia
Major cardiorenal events | about 2 years
  Time to first occurrence of the composite of major adverse cardiorenal events (MACER) as defined as all-cause mortality, stroke, non-fatal myocardial infarction, heart failure events including hospitalization for CHF or urgent CHF treatment, sustained (for at least 3 months) 40% decline in eGFR, or allograft failure as defined by chronic dialysis, re-transplantation, or persistent eGFR <15mL/min/1.73m2)
Acute Graft Dysfunction | about 2 years
  The cumulative incidence of >15% elevation in serum creatinine for more than 4 weeks from the baseline defined prior to treatment.
Volume Depletion | about 2 years
  The cumulative incidence of grade 3 volume depletion.
Acute Cellular Rejection | about 2 years
  The cumulative incidence of acute rejection biopsy proven using 2017 criteria:
  Type IA Moderate tubulitis and at least moderate interstitial inflammation t2i2 or t2i3 Type IB Severe tubulitis and at least moderate interstitial inflammation t3i2 or t3i3 Type IIA Mild to moderate intimal arteritis v1 Type IIB Severe intimal arteritis (> 25% of the luminal area) v2 Type III Transmural' arteritis and/or fibrinoid necrosis v3 Borderline: no intimal arteritis is present, t>0 and i1 or i2/i3 and t1
Amputation and foot ulceration | About 2 years
  The cumulative incidence of Grade 3 foot ulceration and/or need for amputation.
Proteinuria | 12 and 24 months
  Spot Urine Protein/creatinine ratio
Allograft Biopsy | about 2 years
  Time to incidence of a decline in eGFR sufficient to trigger a clinical decision for an allograft biopsy
MACER | about 2 years
  Time to first occurrence of individual component of the MACER secondary outcome
Death | about 2 years
  Time to the occurrence of cardiovascular death
Acute graft dysfunction | About 2 years
  Time to acute kidney injury as defined as a >15% change in eGFR from baseline
Slope of kidney function | over 2 years
  Serum creatinine measured in mg/dL for all participants prior to treatment, at month 6, month 12 and month 24 of treatment.
Glycemic Control | over 2 years
  Changes in Hemoglobin A1C over time of treatment
Body Weight | over 2 years
  Change in body weight over time of treatment
Blood Pressure | over 2 years
  Change in blood pressure measured in mmHg over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Roslyn B Mannon, MD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (5):
- United States (5):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No